CLINICAL TRIAL: NCT00277095
Title: Clinical Investigation of the ProACT Adjustable Continence Therapy for Treatment of Post-Prostatectomy Stress Urinary Incontinence
Brief Title: ProACT Therapy for the Treatment of Stress Urinary Incontinence in Males
Acronym: ProACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uromedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM02
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-04

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ProACT (Adjustable Continence Therapy) (Experimental): Implantation with ProACT (Adjustable Continence Therapy), Single Arm
  Interventions: Device: ProACT (Adjustable Continence Therapy)

INTERVENTIONS:
Device: ProACT (Adjustable Continence Therapy) — Implantable device to reduce urinary stress incontinence
  Other Names: ProACT,Adjustable Incontinence therapy for Males

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of a minimally invasive surgical procedure in up to 109 male patients. The ProACT device is designed to treat men who have stress urinary incontinence arising from intrinsic sphincter deficiency following an operation performed on the prostate for cancer or for benign prostatic hyperplasia. Two adjustable balloons (one on each side of the urethra) are implanted to treat urinary stress incontinence.

The results will be analyzed to demonstrate the effects of the device as well as its associated risks. Therapeutic success will be based on whether patients demonstrate at least a 50% reduction in pad weight at 18 months follow-up compared to the pad weight results at baseline.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized multi-center investigation. Multiple measurements using 24 hour pad weight and pad count, validated questionnaires, voiding diaries will be used to evaluate the achievement of the study objectives. Subjects will be followed for a minimum of 18 months following implantation. Subjects will be requested to continue annual follow-ups through the FDA approval.

The purpose of the study is to evaluate the safety and effectiveness of a minimally invasive surgical procedure in up to 109 male patients. The ProACT device is designed to treat men who have stress urinary incontinence arising from intrinsic sphincter deficiency following an operation performed on the prostate for cancer or for benign prostatic hyperplasia. Two adjustable balloons (one on each side of the urethra) are implanted to treat urinary stress incontinence.

The results will be analyzed to demonstrate the effects of the device as well as its associated risks. Therapeutic success will be based on whether patients demonstrate at least a 50% reduction in pad weight at 18 months follow-up compared to the pad weight results at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Undergone either a radical prostatectomy, transurethral resection of the prostate or other prostate surgery at least 12 months prior without radiation therapy
* Demonstrate primary stress urinary incontinence
* Male subjects at least 45 years of age
* Willing and able to undergo surgical implantation of the ProACT devices
* Willing and able to comply with the follow-up requirements
* Willing and able to forego any other surgical urinary incontinence treatments while participating in the study
* Willing and able to sign the informed consent
* Positive 24 hour pad weight tests (greater than or equal to 8 gram pad weight increase demonstrated in two 24-hour pad weight tests)
* Experiences at least 3 incontinence episodes per day during two baseline voiding diaries.
* Negative Urine culture
* No recurrent stricture at the anastamosis
* No known urogenital malignancy other than previously treated prostate cancer
* Physician determines subject to be suitable surgical candidate

Exclusion Criteria:

* Primarily Urge incontinence
* Detrusor instability or over-activity
* Residual volume greater that 100 ml or greater than 25% of the total bladder capacity after voiding.
* Subject has/had or is suspected of having bladder cancer
* History of recurrent bladder stones
* Neurogenic bladder that is atonic or has detrusor sphincter dyssynergia
* Known hemophilia or a bleeding disorder
* Abnormal PSA (Prostate Specific Antigen), according to sites laboratory standards, unless further investigation confirms no underlying prostate malignancy.
* Known sever contrast solution allergy
* Has a genitourinary mechanical prosthesis other than previous sling procedure (e.g., Artificial Urinary sphincter, implantable penile prosthesis)
* Has a urethral stricture that prevents passage of an 18 F cystoscope or has had more than one urethrotomy
* Undergone bulking procedure within 6 months of the baseline assessment
* Subject is currently enrolled or plans to enroll in another device or drug clinical trial.
* Subject is currently using an indwelling catheter or condom catheter for treatment of incontinence and is not willing to discontinue use at least 4 weeks prior to baseline assessment.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Cook, Ph.D, Study Director — Uromedica, Inc.
Locations (10):
- United States (7):
  - University of Arizona, Tucson, Arizona
  - Kaiser Permanente-Los Angeles, Los Angeles, California
  - The Pelvic Clinic, Pembroke Pines, Florida
  - Indian River Urology, Vero Beach, Florida
  - Urological Surgeons, Kankakee, Illinois
  - Metro Urology, Saint Paul, Minnesota
  - Kansas City Urology Care, Kansas City, Missouri
- Canada (2):
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - CHUS-Fleurimont, Fleurimont, Quebec
- Urology Bay of Plenty (formerly Promed Urology), Tauranga, New Zealand

REFERENCES:
- See also: ProACT Adjustable Continence for Men Premarket Approval (PMA) 11/24/2015 — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPMA/pma.cfm?id=3425

RESULTS

PARTICIPANT FLOW:
Groups:
- Implantable Device: ProACT Implantable device for treatment of post-prostatectomy stress urinary incontinence in males.
Period: Overall Study
Arm/Group | Implantable Device
Started | 124 (Anatomy of 1 patient did not allow ProACT to be implanted, hence only 123 patients were implanted.)
Completed | 103 (Details of patients who did not complete study are given below.)
Not Completed | 21
Not completed — Death | 2
Not completed — Explanted | 7
Not completed — Lost to Follow-up | 2
Not completed — Missed Follow-up | 9
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- ProACT: Implantable device
Arm/Group | ProACT
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 124
Region of Enrollment [Number; unit: participants]
  United States | 68
  Canada | 44
  New Zealand | 12

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: Demonstrate the Efficacy of the ProACT Device in Reducing Incontinence as Measured by the 24-hour Pad Weight at 18 Months Compared to Baseline. A Subject is a Success if he Demonstrates a 50% Reduction.
Description: The percentage of participants with 50% reduction in pad weight.
Time Frame: 18 month follow-up
Population: As followed analysis of all patients who were treated and reached the 18 month follow-up visit
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Urine Loss ( in Grams): 24 hour pad weight(in grams) demonstrating 50% reduction in urine loss (in grams)over 18th month
Arm/Group | Urine Loss ( in Grams)
Number analyzed (Participants) | 99
percentage of patients | 60.6 [50 to 70]

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | ProACT
Serious Adverse Events (participants affected / at risk) | 4/124
Other Adverse Events (participants affected / at risk) | 112/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProACT (N=124)
CVA (Vascular disorders) | 1 (1)
Low Heart Rate (Cardiac disorders) | 1 (1)
Ulcerative Colitis (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProACT (N=124)
Other Genitourinary (Renal and urinary disorders) | 46 (79)
Other Non Genitourinary (General disorders) | 40 (54)
Pain Genitourinary (Renal and urinary disorders) | 35 (47)
Worsening Incontinence (Renal and urinary disorders) | 35 (37)
Balloon Migration (Investigations) | 21 (30)
Infection, Urinary Tract (Renal and urinary disorders) | 20 (23)
Retention (Renal and urinary disorders) | 18 (23)
Perforation During Implant (Investigations) | 17 (20)
Dermotologic (Skin and subcutaneous tissue disorders) | 13 (15)
Gastrointestinal Condition (Gastrointestinal disorders) | 13 (14)
Oncological/hematologic Condition (Blood and lymphatic system disorders) | 13 (13)
Device Failure, Leakage (Investigations) | 10 (10)
Infection, Genitourinary (Infections and infestations) | 9 (11)
Balloon Erosion (Investigations) | 8 (8)
Pain, nongenitourinary (General disorders) | 8 (9)
Cardiac Condition (Cardiac disorders) | 7 (8)
Device Failure, other (Investigations) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No